CLINICAL TRIAL: NCT04007055
Title: The Value of Screening for "High on Treatment Platelet Reactivity" in Patients Undergoing Lower Extremity Arterial Endovascular Interventions
Brief Title: The Value of Screening for HPR in Patients Undergoing Lower Extremity Arterial Endovascular Interventions
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Marissa Jarosinski (Other)
Responsible Party: Sponsor-Investigator, Marissa Jarosinski, Resident in Vascular Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY19030453
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Artery Disease; Clopidogrel, Poor Metabolism of; Peripheral Vascular Disease; Artery Disease; Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Peripheral Arterial Occlusive Disease 1 | interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: screening/treating for HPR (Experimental): Participants randomized to this arm will be screened and treated for HPR. Pharmacogenetics testing for CYP2C19 polymorphisms will be collected, stored, and analyzed at study completion.
  Interventions: Diagnostic Test: Point of care screening for HPR; Drug: Ticagrelor 90mg
- Control: guideline based therapy (No Intervention): Participants randomized to this arm will receive usual care without screening for HPR. Pharmacogenetics testing for CYP2C19 polymorphisms will be collected, stored, and analyzed at study completion.

INTERVENTIONS:
Diagnostic Test: Point of care screening for HPR — HPR testing using VerifyNow testing system. HPR is defined platelet reactivity units are greater than 234
  Arms: Experimental: screening/treating for HPR
Drug: Ticagrelor 90mg — Participants who test positive for HPR will be prescribed ticagrelor 90mg twice daily instead of standard therapy with clopidogrel 75mg daily
  Arms: Experimental: screening/treating for HPR

SUMMARY:
This is a randomized controlled trial designed to evaluate the role of screening for and intervening on patients with high on treatment platelet reactivity undergoing lower extremity arterial endovascular interventions.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects millions of people worldwide. Management of PAD has evolved from open surgery to an endovascular first approach leading to increased volume of endovascular interventions. Endovascular femoropopliteal intervention has emerged as a standard treatment for symptomatic PAD with acceptable patency rates.

Histologic observation of bare metal stents with early failure shows association with platelet rich thrombus, high counts of platelets, and neutrophils associated with stent struts. Additionally, high inflation pressures associated with balloon angioplasty often causes local tissue damage leading to platelet activation. These findings led to studies targeting platelet activation following endovascular treatment showing improved outcomes in patients receiving stronger platelet inhibition.

The current standard of care is prescription of dual antiplatelet therapy (DAPT) for femoropopliteal angioplasty or stenting. DAPT is active use of any two antiplatelet agents, often low dose aspirin plus P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel). There is improved stent patency and reduced adverse cardiovascular events in patients taking DAPT versus aspirin monotherapy.

Clopidogrel is the most common additional antiplatelet agent prescribed, but 4-65% of patients taking clopidogrel fail to achieve clinically expected platelet inhibition. This persistent platelet reactivity despite compliant antiplatelet use is commonly referred to as high on-treatment platelet reactivity (HPR), and increases risk of endovascular intervention failure and associated adverse clinical events in these patients. Clopidogrel is a pro-drug metabolized by CYP2C19 enzyme into its active form. Failure to respond appropriately to clopidogrel is largely due to genetic polymorphisms within CYP2C19 enzyme resulting in variable metabolization of clopidogrel into the active metabolite.

Alternative antiplatelet medications can overcome HPR through different metabolic pathways, but unfortunately at a significantly higher cost. Of these, ticagrelor is often used to overcome HPR for patients taking clopidogrel with favorable outcomes. However, regional cost for ticagrelor is $352.50 compared to $1.96 for clopidogrel. Cost and bleeding concerns among providers have prevented widespread use. Overall, there is paucity of evidence looking at HPR and lower extremity arterial endovascular interventions without consensus or guidelines on how to address this problem. Thus, the investigators propose an unblinded, randomized controlled trial in patients having femoropopliteal angioplasty or stenting comparing two strategies: 1. testing and treating for HPR versus 2. guideline based therapy without testing for HPR.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease
* Planned angioplasty or stenting of superficial femoral artery or popliteal artery.

Exclusion Criteria:

* Patients treated on an emergency basis
* Planned intervention on prior site of open surgical intervention (autogenous or autologous bypass, endarterectomy, or patch angioplasty)
* Planned intervention at site exclusive of superficial femoral artery or popliteal artery
* Planned re-stenting at site of prior stent placement
* Planned re-angioplasty at site of prior angioplasty
* Known inability to tolerate antiplatelet regimen before enrollment
* Patients who plan on receiving follow up care outside the University of Pittsburgh Medical Center
* Current use of prasugrel or ticlopidine
* Current use of oral anticoagulation medication
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with primary patency | one year from intervention
  primary patency is freedom from re-intervention, freedom from complete vessel occlusion, freedom from >50% restenosis with duplex ultrasound or freedom from >70% restenosis with computed tomography angiography

SECONDARY OUTCOMES:
proportion of participants with amputation | one year from intervention
  Freedom from new amputation on the lower extremity intervened on during study
Correlation of HPR testing results | after study completion
  Correlation of HPR results between VerifyNow and CYP2C19 pharmacogenetics testing
Major adverse cardiovascular events | one year from intervention
  Any new stroke, myocardial infarction, death during study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No